CLINICAL TRIAL: NCT05455320
Title: A Phase 3 Randomized Study Comparing Talquetamab SC in Combination With Daratumumab SC and Pomalidomide (Tal-DP) or Talquetamab SC in Combination With Daratumumab SC (Tal-D) Versus Daratumumab SC, Pomalidomide and Dexamethasone (DPd), in Participants With Relapsed or Refractory Multiple Myeloma Who Have Received at Least 1 Prior Line of Therapy
Brief Title: A Study Comparing Talquetamab in Combination With Daratumumab or in Combination With Daratumumab and Pomalidomide Versus Daratumumab in Combination With Pomalidomide and Dexamethasone in Participants With Multiple Myeloma That Returns After Treatment or is Resistant to Treatment
Acronym: MonumenTAL-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109082; 64407564MMY3002 (Other: Janssen Research & Development, LLC); 2021-000202-22 (EudraCT Number); 2021-000202-22-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05757973 (Approved for marketing)
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — talquetamab; daratumumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Talquetamab Subcutaneous (SC) in Combination With Daratumumab SC and Pomalidomide (Tal-DP) (Experimental): Participants will receive talquetamab and daratumumab as SC injections; pomalidomide will be self-administered as a single dose orally; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: Talquetamab; Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone
- Arm B: Daratumumab in Combination With Pomalidomide and Dexamethasone (DPd) (Experimental): Participants will receive daratumumab as SC injection; pomalidomide will be self-administered as a single dose orally; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone
- Arm C: Talquetamab SC in Combination With Daratumumab SC (Tal-D) (Experimental): Participants will receive talquetamab and daratumumab as SC injection; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: Talquetamab; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564
  Arms: Arm A: Talquetamab Subcutaneous (SC) in Combination With Daratumumab SC and Pomalidomide (Tal-DP); Arm C: Talquetamab SC in Combination With Daratumumab SC (Tal-D)
Drug: Daratumumab — Daratumumab will be administered subcutaneously.
Drug: Pomalidomide — Pomalidomide will be administered orally.
  Arms: Arm A: Talquetamab Subcutaneous (SC) in Combination With Daratumumab SC and Pomalidomide (Tal-DP); Arm B: Daratumumab in Combination With Pomalidomide and Dexamethasone (DPd)
Drug: Dexamethasone — Dexamethasone will be administered orally or intravenously.

SUMMARY:
The purpose of the study is to compare the efficacy of talquetamab subcutaneous(ly) (SC) in combination with daratumumab SC and pomalidomide (Tal-DP) and talquetamab SC in combination with daratumumab SC (Tal-D), respectively, with daratumumab SC in combination with pomalidomide and dexamethasone (DPd).

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma as defined: a) Multiple myeloma diagnosis according to the International Myeloma Working Group (IMWG) diagnostic criteria and b) Measurable disease at screening as defined by any of the following: i) Serum M-protein level greater than or equal to (>=) 0.5 grams per deciliter (g/dL) (central laboratory); ii) Urine M-protein level >= 200 milligram (mg) per 24 hours (central laboratory); iii) Light chain multiple myeloma without measurable M-protein in the serum or the urine: serum immunoglobulin free light chain >= 10 milligram per deciliter (mg/dL) (central laboratory), and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Relapsed or refractory disease as defined by: i) Relapsed disease is defined as an initial response to prior treatment, followed by confirmed progressive disease by IMWG criteria greater than (>) 60 days after cessation of treatment; ii) Refractory disease is defined as less than (<) 25 percent (%) reduction in monoclonal paraprotein (M-protein) or confirmed progressive disease by IMWG criteria during previous treatment or less than or equal to (<=) 60 days after cessation of treatment
* Received at least 1 prior line of antimyeloma therapy including a proteasome inhibitor (PI) and lenalidomide. Participants who have received only 1 prior line of antimyeloma therapy must be considered lenalidomide-refractory (that is, have demonstrated progressive disease by IMWG criteria on or within 60 days of completion of lenalidomide-containing regimen). Participants who have received >=2 prior lines of antimyeloma therapy must be considered lenalidomide exposed
* Documented evidence of progressive disease based on investigator's determination of response by the IMWG criteria on or after their last regimen
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 at screening and immediately prior to the start of administration of study treatment

Exclusion Criteria:

* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to study drug excipients
* Disease is considered refractory to an anti-cluster of differentiation 38 (CD38) monoclonal antibody as defined per IMWG consensus guidelines (progression during treatment or within 60 days of completing therapy with an anti-CD38 monoclonal antibody)
* Received prior pomalidomide therapy
* A maximum cumulative dose of corticosteroids to >=140 milligrams (mg) of prednisone or equivalent within 14-day period before the first dose of study drug
* Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Plasma cell leukemia (per IMWG criteria) at the time of screening, Waldenström's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes (POEMS syndrome), or primary amyloid light chain amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 6 years 6 months
  PFS is defined as time from the date of randomization to the first documentation of disease progression, or death due to any cause, whichever is reported first.

SECONDARY OUTCOMES:
Overall Response (Partial Response [PR] or Better) | Up to 6 years 6 months
  Overall response (PR or better) is defined as percentage of participants who have a PR or better per International Myeloma Working Group (IMWG) criteria.
Very Good Partial Response (VGPR) or Better Rate | Up to 6 years 6 months
  VGPR or better rate is defined as the percentage of participants who achieve a VGPR or better according to IMWG response criteria.
Complete Response (CR) or Better Rate | Up to 6 years 6 months
  CR or better rate is defined as the percentage of participants who achieve CR or better according to IMWG response criteria.
Overall Minimal Residual Disease (MRD) Negative CR | Up to 6 years 6 months
  MRD-negative CR is defined as proportion of participants with CR or stringent CR who achieve MRD negativity at a threshold of 10^-5 at any timepoint after the first dose of study drug and before disease progression or start of subsequent antimyeloma therapy.
Overall Survival (OS) | Up to 6 years 6 months
  OS is defined as the time from the date of randomization to the date of the participant's death.
Progression-free Survival on Next-line Therapy (PFS2) | Up to 6 years 6 months
  PFS2 is defined as the time interval between the date of randomization and date of event, which is defined as progressive disease as assessed by investigator on the first subsequent line of antimyeloma therapy, or death from any cause, whichever occurs first.
Time to Next Therapy (TTNT) | Up to 6 years 6 months
  TTNT is defined as the time from randomization to the start of subsequent antimyeloma treatment.
Number of Participants with Adverse Events (AEs) | Up to 6 years 6 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 6 years 6 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).
Serum Concentrations of Talquetamab | Up to 6 years 6 months
  Serum concentrations of talquetamab will be reported.
Serum Concentrations of Daratumumab | Up to 6 years 6 months
  Serum concentrations of daratumumab will be reported.
Number of Participants with Presence of Anti-Drug Antibodies (ADAs) to Talquetamab | Up to 6 years 6 months
  Number of participants with presence ADAs to talquetamab will be reported.
Number of Participants With Presence of Anti-Drug Antibodies (ADAs) to Daratumumab | Up to 6 years 6 months
  Number of participants with presence of ADAs to daratumumab will be reported.
Time to Worsening in Symptoms, Functioning, and Overall Health-Related Quality of Life (HRQoL) as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) | Up to 6 years 6 months
  The MySIm-Q is a disease-specific PRO assessment complementary to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item (EORTC-QLQ-C30).
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by PROMIS Short Form Version 2.0 -Physical Functioning 8c | Up to 6 years 6 months
  The Patient-reported Outcomes Measurement Information System (PROMIS) Short Form Version 2.0 -Physical Function 8c is an 8-item fixed--length short form derived from the PROMIS Physical Function item bank.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by EORTC-QLQ-C30 | Up to 6 years 6 months
  Time to worsening in symptoms, functioning, and HRQoL as assessed by EORTC-QLQ-C30 will be reported.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by PRO-CTCAE | Up to 6 years 6 months
  The National Cancer Institute's (NCI) PRO-CTCAE is an item library of common AEs experienced by people with cancer that are appropriate for self-reporting of treatment tolerability.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | Up to 6 years 6 months
  The EQ-5D-5L is a generic measure of health status. For purposes of this study, the EQ-5D-5L will be used to generate utility scores for use in cost-effectiveness analyses.
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by Patient Global Impression - Severity (PGI-S) | Up to 6 years 6 months
  The PGI-S will be used as an anchor, external criterion, to determine meaningful change in scores for the MySIm-Q and PROMIS SF PF 8c in this population.
Change From Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) | Baseline up to 6 years 6 months
  The MySIm-Q is a disease-specific PRO assessment complementary to the EORTC-QLQ-C30.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by PROMIS Short Form Version 2.0 -Physical Functioning 8c | Baseline up to 6 years 6 months
  The Patient-reported Outcomes Measurement Information System (PROMIS) Short Form Version 2.0 -Physical Function 8c is an 8-item fixed-length short form derived from the PROMIS Physical Function item bank.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by EORTC-QLQ-C30 | Baseline up to 6 years 6 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by EORTC-QLQ-C30 will be reported.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by PRO-CTCAE | Baseline up to 6 years 6 months
  The National Cancer Institute's (NCI) PRO-CTCAE is an item library of common AEs experienced by people with cancer that are appropriate for self-reporting of treatment tolerability.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | Baseline up to 6 years 6 months
  The EQ-5D-5L is a generic measure of health status. For purposes of this study, the EQ-5D-5L will be used to generate utility scores for use in cost-effectiveness analyses.
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by Patient Global Impression - Severity (PGI-S) | Baseline up to 6 years 6 months
  The PGI-S will be used as an anchor, external criterion, to determine meaningful change in scores for the MySIm-Q and PROMIS SF PF 8c in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (216):
- United States (40):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Norwalk Hospital-oncology, Norwalk, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - University of Miami Health System, Miami, Florida
  - University Of Illinois, Chicago, Illinois
  - University of Kansas, Westwood, Kansas
  - Tulane University Hospital & Clinics, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School Of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Health, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio
  - OhioHealth, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research Treatment Center, Lubbock, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (6):
  - UZ Brussel, Brussels
  - UZA, Edegem
  - Virga Jessa Ziekenhuis, Hasselt
  - CHC MontLegia, Liège
  - Clinique Saint Pierre, Ottignies
  - UCL Mont Godinne, Yvoir
- Brazil (17):
  - Fundacao Pio XII, Barretos
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Hospitais Integradaos da Gavea S/A - DF Star, Brasília
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Hospital Paulistano, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Clinica Sao Germano, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- China (19):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The second Xiangya Hospital of Central South University, Changsha
  - Beijing Chaoyang Hospital, Chaoyang District
  - Sichuan Academy of Medical Science Sichuan Provincial People's Hospital, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat Sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Tongji Hospital of Tongji University, Shanghai
  - Shanghai Fourth People s Hospital, Shanghai
  - Peking University Shenzhen Hospital, Shenzhen
  - First Affiliated Hospital SooChow University, Suzhou
  - Tianjin cancer hospital, Tianjin
  - Institute of Hematology & Blood Disease Hospital Chinese Academy of Medical Science, Tianjin
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze - I. interni klinika - klinika hematologie, Prague
- France (9):
  - APHP - Hopital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - Centre Leon Berard, Lyon
  - CHU de Montpellier - Hopital Saint-Eloi, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - CHU HOPITAL DE L'ARCHET - Hematology, Nice
  - CHU Hopital Saint Antoine, Paris
  - CHRU - Hôpital du Haut Lévêque - Centre François Magendie, Pessac
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- Germany (7):
  - Charite Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg Universität, Mainz
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - Alexandra General Hospital of Athens, Athens Attica
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - G Papanikolaou Hospital of Thessaloniki, Thessalonikis
- Israel (12):
  - Ha'Emek Medical Center, Afula
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Beilinson medical center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
  - Sourasky (Ichilov) Medical Center, Tel Aviv
- Italy (14):
  - A.O. Universitaria Ospedali Riuniti di Ancona, Ancona
  - Policlinico di Bari, Bari
  - Azienda Ospedaliera Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - PO G.Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Ospedale Villa Sofia-Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - Presidio Ospedaliero Santo Spirito in Sassia, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O.U. Città della Salute e della Scienza, Torino
- Japan (21):
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - Fukuoka University Hospital, Fukuoka
  - Ogaki Municipal Hospital, Gifu
  - Gunma University Hospital, Gunma
  - Kansai Medical University Hospital, Hirakata
  - Hyogo Medical University Hospital, Hyôgo
  - Japanese Red Cross Society Himeji Hospital, Hyōgo
  - Shonan Kamakura General Hospital, Kamakura-shi
  - National Cancer Center Hospital East, Kashiwa
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Kumamoto University Hospital, Kumamoto
  - Kyoto Kuramaguchi Medical Center, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Niigata Cancer Center Hospital, Niigata
  - National Hospital Organization Hiroshima-Nishi Medical Center, Ōtake
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Iwate Medical University Hospital, Shiwa-gun
  - The University of Osaka Hospital, Suita
  - The Cancer Institute Hospital of JFCR, Tokyo
- Netherlands (3):
  - Albert Schweitzer ziekenhuis-lokatie Dordwijk, Dordrecht
  - Maxima Medisch Centrum, Eindhoven
  - Erasmus MC, Rotterdam
- Poland (11):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Szpital Kliniczny MSWiA z Warminsko Mazurskim Centrum Onkologii w Olsztynie Oddzial Hematologii, Olsztyn
  - Uniwersytecki Szpital Kliniczny Nr 1 PUM im prof Tadeusza Sokolowskiego w Szczecinie, Szczecin
  - Wojewodzki Szpital Zespolony im L Rydygiera w Toruniu, Torun
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- South Korea (10):
  - Dong-A University Hospital, Busan
  - National Cancer Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (16):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Virgen de La Arrixaca, El Palmar
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. de Leon, León
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. de Canarias, San Cristóbal de La Laguna
  - Hosp. Univ. Dr. Peset, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (9):
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Hematology Unit, Ankara
  - Ankara University Medical Faculty, Ankara
  - Liv Hospital Ankara, Ankara
  - Antalya Training And Research Hospital, Antalya
  - Medipol Mega University Hospital, Istabul
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ondokuz Mayis University, Samsun
- United Kingdom (8):
  - Blackpool Victoria Hospital, Blackpool
  - Ninewells Hospital & Medical School, Dundee
  - Hammersmith Hospital, London
  - Newcastle Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Marsden Hospital, Sutton
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- See also: Click here to learn more about the 64407564MMY3002 (MonumenTAL-3) trial — https://sparkcures.com/trial/1328/nct05455320?utm_source=ctgov&utm_medium=organic&utm_campaign=monumental3